CLINICAL TRIAL: NCT03758794
Title: Knowledge and Attitude of Dental Interns on Child Abuse After Implementation of Two Educational Modules: A Randomized Control Trial
Brief Title: Knowledge and Attitude of Dental Interns on Child Abuse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maria Nabil Leithy Dawood, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: nld201151
Record Dates: First submitted 2018-11-25; First posted 2018-11-29 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Child Abuse

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interactive lecture module (Active Comparator): interactive lecture
  Interventions: Other: interactive lecture
- online educational module (Active Comparator): online educational using a special link
  Interventions: Other: online education

INTERVENTIONS:
Other: interactive lecture — an interactive lecture will be given to a group of dental interns students on child abuse recognition and reporting
  Arms: interactive lecture module
Other: online education — an online educational module will be sent to a group of dental interns students on child abuse recognition and reporting
  Arms: online educational module

SUMMARY:
1. Knowledge and attitude of dental interns of the pediatric dental department regarding child abuse recognition and reporting will be assessed 2 times before and after attending one of 2 learning modules ( interactive lecture or online module ) assessment through a questionnaire
2. assessment of the learning experience through a written questionnaire

DETAILED DESCRIPTION:
1. An introduction with the aim of the study will be given to all the interns of the pediatric dentistry department, Faculty of Dentistry, Cairo University during a regular scheduled seminar.
2. All interns willing to join the study will be asked to sign an informed consent.
3. A pre-test questionnaire on recognition and reporting of child abuse will be given to the participants
4. The participants will be randomly allocated to 2 study groups Online Group: (this group will receive the educational material through an online educational module ) Lecture Group: (this group will receive the educational material through an interactive lecture based educational module )
5. A post-test same as the pre-test will be used to assess the change in knowledge and attitude regarding child abuse recognition and reporting after the completion of the assigned educational module.
6. All participants that attended both educational modules will be asked to answer a small questionnaire about their perceptions regarding the learning experience.

ELIGIBILITY:
Inclusion Criteria:

* Dental Interns enrolled in the Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Cairo University
* Participants of both genders
* Graduates of any dental school in Egypt

Exclusion Criteria:

* Participants who refused to sign the consent
* Participants who won't be able to have online access to the material

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Questionnaire on Knowledge and Attitude of child abuse | 2 questionnaires each for 15 minutes before and after the learning module
  assess the change in knowledge and attitude of dental interns regarding child abuse before and after the educational module assigned to the group same questionnaire will be given pre and post the educational module the questionnaire will include 25 multiple choice questions each question will score 4 with the total questionnaire out of 100 . the questionnaire that will score 75 or less will be considered failed

SECONDARY OUTCOMES:
Questionnaire on Perception of the learning experience | A 10 minutes written questionnaire
  assessment of the dental interns' perception of the educational module the questionnaire will include 7 questions about how strongly or not they preferred the educational module administrated or not evaluation of the answers and comparison between both educational modules according to the % of agreement on each module each question will be analysed with comparison between the % of interns who strongly agree, agree, neutral, disagree or strongly disagree

REFERENCES:
- [Derived] Walsh K, Eggins E, Hine L, Mathews B, Kenny MC, Howard S, Ayling N, Dallaston E, Pink E, Vagenas D. Child protection training for professionals to improve reporting of child abuse and neglect. Cochrane Database Syst Rev. 2022 Jul 5;7(7):CD011775. doi: 10.1002/14651858.CD011775.pub2. PMID 35788913